CLINICAL TRIAL: NCT01538563
Title: Phase I Dose Escalation Study of ON 01910.Na by 24 Hour Continuous Infusion Per Week in Patients With Advanced Cancer
Brief Title: Safety of 24-Hour Infusion of ON 01910.Na in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Onconova 04-03
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Solid Tumors; Advanced Cancer; Cancer; Neoplasms
Keywords: ON 01910.Na; rigosertib sodium; rogosertib
MeSH Terms: conditions — Neoplasms | interventions — ON 01910

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: rigosertib sodium — Patients will receive escalating doses of ON 01910.Na (250 mg/m2 to 4450 mg/m2) intravenously by 24 hour continuous infusion once every week (3 weeks per cycle), until evidence of disease progression, intolerable adverse events, or withdrawal of patient consent.
  Other Names: ON 01910.Na Concentrate; ON 01910.Na; rigosertib

SUMMARY:
The primary purpose of this study is to determine the highest dose of ON 01910.Na that can be safely given as an intravenous infusion over 24 hours once a week in a 3-week cycle to patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is an open-label, dose-escalating Phase I study of ON 01910.Na in patients with advanced cancers, who have satisfied the inclusion/exclusion criteria enumerated in this protocol. Patients will receive ON 01910.Na intravenously by 24 hour continuous infusion once every week (3 weeks per cycle), until evidence of disease progression, intolerable adverse events, or withdrawal of patient consent. Safety monitoring will be done for at least 3 weeks before escalation to the next dose level. As of Amendment 7, up to 6 patients with gynecological malignancies will be enrolled at the 2400 mg/m2 dose level to determine the appropriateness of this dose as the Recommended Phase Two Dose (RPTD).

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically confirmed solid tumor (leukemias and lymphomas excluded) malignancy that is incurable and for which standard (FDA approved or established standard clinical practice), curative, or palliative measures do not exist or are no longer effective.
* Patients with disease amenable to sequential biopsies will be requested to undergo two tumor biopsies and two normal skin biopsies, but patients may decline and still be eligible for enrollment during this escalation stage.
* At least 3 weeks since the last dose of other potentially myelosuppressive treatment (at least 6 weeks since last dose of nitrosoureas or mitomycin C) and recovery from manifestations of reversible drug toxicity (alopecia, stable residual neuropathy, and residual hand and foot syndrome are excluded). Patients with prior doxorubicin chemotherapy must have total cumulative dose of no more than 450 mg/m2.
* Patients with prior radiotherapy are eligible provided a minimum of 4 weeks have passed and the maximal area of hematopoietic active bone marrow treated was less than 25%.
* ECOG performance status ≤2.
* Patients must have nearly normal organ and marrow function as defined below:
* Hgb > 9 gm/dl (must not require transfusional support but erythropoietin therapy is permitted)
* WBC > 4,000 per microliter
* Absolute neutrophil count > 1,500 per microliter
* Platelets ≥ 100,000 per microliter
* Total bilirubin within 1.5 times institutional upper normal limit
* AST(SGOT)/ALT(SGPT) ≤ 2.5 x institutional upper normal limit. (If liver function abnormalities are due to metastatic disease, patients are eligible provided the transaminases are < 5 times institutional upper normal limit. Patients with primary liver disease with these parameters will be ineligible.)
* Serum creatinine within normal institutional limits or estimated creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry.
* Ability to understand and the willingness to sign a written informed consent document.
* All ethnic groups are eligible for this trial.

Inclusion Criteria - Dose Confirmation Phase Same inclusion criteria as in the Dose Escalation phase described above, except Patients must have an ECOG performance of 0 or 1.

Exclusion Criteria:

* Recent major surgery (within the past 14 days), chemotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) or radiotherapy within 4 weeks prior to entering the study, or those who have not recovered from adverse events (except alopecia, stable residual neuropathy, and residual hand and foot syndrome) due to previously administered agents.
* Patients may not be on any other investigational agents or concurrent chemotherapy, radiotherapy, hormonal treatments, bone marrow transplantation, or immunotherapy. Patients who have previously had a Bone Marrow Transplant are excluded from this study.
* Known brain metastases, except brain metastases that have been previously removed or irradiated and currently have no clinical impact.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ON 01910.Na.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, bleeding, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and nursing women are excluded.
* HIV-positive patients receiving combination anti-retroviral therapy are excluded.
* Ascites requiring active medical management including paracentesis, peripheral bilateral edema, hyponatremia (serum sodium value less than 134 Meq/L).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-06; Primary Completion 2010-07 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Number of dose limiting toxicities (DLTs) | 21 days after first administration of ON 01910.Na
  DLTs are defined as:
  * Grade 3 non-hematological toxicity other than nausea, vomiting, diarrhea, fever, stomatitis, esophagitis/dysphagia.
  * Recurrent grade 3 toxicity uncontrolled by optimal therapy or Grade 4 nausea, vomiting, diarrhea and fever.
  * Grade 3 stomatitis and/or esophagitis/dysphagia for > 5 days.
  * Grade 4 neutropenia or thrombocytopenia for > 5 days measured at least 2X 2-3 days apart.
  * Neutropenic fever, as defined in Protocol.
  * Failure to recover neutrophils (> 1,500 per microliter) or platelets (>75,000 per microliter) before the next weekly dose.

SECONDARY OUTCOMES:
Number of Adverse Events (AEs) | 30 days after last infusion of study drug
  All AEs (except Grade 1 and 2 laboratories abnormalities that do not require an intervention) are recorded in Case Report Forms and source documentation.
Severity of Adverse Events (AEs) | 30 days after last infusion of study drug
  Severity of AEs are determined according to Common Terminology Criteria for Adverse Events (Version 3.0)
Relationship of Adverse Events (AEs) to Study Treatment | 30 days after last infusion of study drug
  Relationship assessed as Not related, Unlikely, Possibly, Probably, or, Definitely according to Guidance in Appendix II of Protocol.
Concentration of ON 01910.Na in plasma versus time | Up to 48 hours after infusion of study drug during Week 1 in Cycles 1 and 2
  Blood samples will be collected at following time points: Pre-dose; 1 h after start of infusion; 3 h; 6 h; 12 h; 18 h; 24 h; 10 min after end of infusion; 20 min; 30 min; 1 h; 2 h; 4 h; 8 h; 24 h; and, 48 h. Plasma will be prepared from these samples. Concentration of ON 01910.Na will be determined by validated method.
Change in size of target lesions recorded at baseline | 30 days after last infusion of study drug
  The same method of assessment for each identified and recorded lesion will be used at baseline and each follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Sridhar Mani, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein Cancer Center, The Bronx, New York, United States

REFERENCES:
- [Result] Garcia-Manero G, Fenaux P. Comprehensive Analysis of Safety: Rigosertib in 557 Patients with Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML). Blood Dec 2016, 128 (22) 2011; ASH 2016.